CLINICAL TRIAL: NCT05994079
Title: Effect Of High-Intensity Focused Ultrasound On Abdominal Skin Laxity Post Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Hassan Kamel Abdelkader El-Hawary, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 012/003743
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Skin Laxity; Gastrostomy
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high intensity focused ultrasound group (Experimental): This group includes 43 patients who have abdominal skin laxity post sleeve gastrectomy and who will receive high intensity focused ultrasound. patients will receive one session; time of session is 40 minutes.
  Interventions: Device: High intensity focused ultrasound
- medical topical firming creams group (Active Comparator): This group includes 43 patients who have abdominal skin laxity post sleeve gastrectomy and who will receive medical topical firming creams.
  Interventions: Other: topical firming creams

INTERVENTIONS:
Device: High intensity focused ultrasound — Parameters:
  Transducer frequency 7-2-mhz 1.5-9.0-mm focal depth. The pulse duration for each individual exposure ranged from 25 to 40 milliseconds.
  Energy per ultrasound pulse ranged from 1.0 to 1.5 J
  Arms: high intensity focused ultrasound group
Other: topical firming creams — medical topical firming creams
  Arms: medical topical firming creams group

SUMMARY:
The purpose of the study is to evaluate the therapeutic effect of High intensity focused ultrasound in treatment of abdominal skin laxity post sleeve gastrectomy.

DETAILED DESCRIPTION:
Lax skin is a common consequence of bariatric weight loss, and it may require one or more plastic interventions.

This study carried out to investigate the effectiveness of High-intensity focused ultrasound (HIFU) in treatment of abdominal skin laxity post sleeve gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

The subject selection will be according to the following criteria:

* Age range between 30-45 years.
* Female patients will participate in the study.
* All patients will have post sleeve gastrectomy abdominal skin laxity mild to moderate degree according to skin laxity scale Randomized images were evaluated by three clinical specialists for the degree of skin laxity (0-3 scale; 0 = no laxity, 1 = mild, 2 = moderate, 3 = severe).
* All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

The potential participants will be excluded if they meet one of the following criteria:

* Age more than 45 years or less than 30 years.
* Patients have acute viral diseases, acute tuberculosis, mental disorders
* Older people with more extensive photo-aging, severe skin laxity.
* Open skin lesions at the target area.
* Severe or cystic acne.
* Metallic implants in the treatment area.
* Genetic disease
* Skin infectious diseases.
* Sociological diseases.
* Pregnant.

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Assessment othe change in skin laxity | at baseline and after 4 weeks of intervention
  By Investigator Global Aesthetic Improvement Scale (IGAIS).
  * The investigator will take clinical photographs using consistent patient positioning, camera settings (Canon EOS 600D, high-resolution setting, 5760 × 3840 pixels, Canon Inc., Tokyo, Japan), and room lighting.
  * Baseline and post-treatment photographs will randomly displayed, and evaluated by Investigator Global Aesthetic Improvement Scale (IGAIS) scores will be determined using side-by-side comparisons of pretreatment and post 4 weeks of treatment.
  * The scale ranges from 0 to 3 as 0 = No change, 1 = Mild improvement, 2 = Moderate improvement, 3 = Significant improvement.
Assessment the change in abdominal skin laxity | at baseline and after 4 weeks of intervention
  Assessment of abdominal skin laxity by the modified tissue tonometer :
  Mark multiple points to be measured. Include an equivalent normal skin point(s).
  Apply the MTT baseplate directly to the tissue through the holes in the template. Hold MTT vertically, with bubble of spirit level centered. Ensure no extra downward pressure is applied while resting the device on the tissue.
  Record the depression of the plunger in millimeters after 6 seconds. The patient must be able to remain immobile when the MTT is in contact.
  Repeat each point three times with at least 2 minutes' "rest" between attempts. Recalibrate the device to zero on a solid surface between each set of measures.
  To determine longitudinal change in measures, comparison of averaged score for individual points is appropriate and/or analysis of the change of individual sagging points difference from normal skin control point(s).

CONTACTS AND LOCATIONS:
Overall Officials: Rania Elhawary, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic faculty of physical therapy cairo university, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No